CLINICAL TRIAL: NCT05225857
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Absolute Bioavailability, Pharmacokinetics, and Pharmacodynamics of AGA2118 in Men and Postmenopausal Women
Brief Title: A First-in-Human Study Evaluating AGA2118 in Men and Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Angitia Biopharmaceuticals (Industry)
Collaborators: Angitia Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-001
Record Dates: First submitted 2022-01-11; First posted 2022-02-07 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AGA2118 (Experimental): In SAD part, various single doses of AGA2118 will be administered to the participants via either SC injection or IV infusion. The starting dose was 0.3 mg/kg, with sequential escalation up to 15 mg/kg.
  In MAD part, various multiple doses of AGA2118 will be administered every four weeks (Q4W) to the participants via SC injection for 12 weeks. The starting dose was 1 mg/kg, with sequential escalation up to 12 mg/kg.
  Interventions: Drug: AGA2118
- Placebo (Placebo Comparator): In SAD part, a single dose of placebo comparator will be used for each cohort of either SC or IV administration.
  In MAD part, multiple doses of placebo comparator will be used for each cohort of SC administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AGA2118 — Part 1 - SAD study: SAD participants in various cohorts will receive various single dose of AGA2118 via either SC or IV.
  Part 2 - MAD study: MAD participants in various cohorts will receive various multiple doses of AGA2118 Q4W via SC.
  Arms: AGA2118
Drug: Placebo — Part 1 - SAD study: SAD participants in various cohorts will receive a single dose of placebo via either SC or IV.
  Part 2 - MAD study: MAD participants in various cohorts will receive multiple doses of placebo via SC.
  Arms: Placebo

SUMMARY:
The primary objectives of the study are to assess the safety and tolerability of AGA2118 after single subcutaneous or intravenous administration in healthy men and postmenopausal women and to assess the safety and tolerability of AGA2118 after multiple subcutaneous administrations in men and postmenopausal women.

DETAILED DESCRIPTION:
This is a Phase I, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Absolute Bioavailability, Pharmacokinetics, and Pharmacodynamics of AGA2118 in Men and Postmenopausal Women.

The study consists of the single ascending dose (SAD) part and the multiple ascending dose (MAD) part. In the SAD part, up to 56 healthy men and postmenopausal women will be sequentially enrolled to receive a single subcutaneous (SC) dose of AGA2118 or a single intravenous (IV) dose of AGA2118 or placebo. In the MAD part, up to 32 healthy men and postmenopausal women will be sequentially enrolled in various dose cohorts to receive multiple SC doses every 4 weeks of AGA2118 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men ≥ 30 and ≤ 65 years of age or postmenopausal women ≥ 45 and ≤ 65 years of age for SAD and MAD;
2. BMI ≥ 18.5 and ≤ 32 kg/m^2 (for SAD and MAD).
3. Generally healthy (as assessed by the investigator).
4. Nonsmokers, or light smokers, defined as ≤ 3 cigarettes/day (or equivalent) (for SAD and MAD).
5. Able and willing to correctly and independently complete all study procedures and able to read, understand, and provide written informed consent after the nature of the study has been fully explained and must be willing to comply with all study requirements and procedures (for SAD and MAD).
6. A male who is sterile or agrees to the following during the Treatment Period and for at least 6 months after the final dose of investigational product

   * Refrain from donating fresh unwashed semen

Plus, either

* Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent

OR

* Must agree to use contraception as detailed below

  * Agree to use a male condom plus a female partner to use a highly effective method of contraception with a woman of childbearing potential who is not currently pregnant
  * Agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person

Exclusion Criteria:

1. A bone fracture within 6 months (for SAD only).
2. Previous exposure to AGA2118 (for MAD only).
3. Any condition that would affect bone metabolism or has a history of low energy fractures as documented in medical history (for MAD only).
4. Administration of the any medications that known to affect bone metabolism within 6 months of Day 1 unless otherwise specified (for SAD and MAD).
5. Human immunodeficiency virus (HIV) infection (for SAD and MAD).
6. Active chronic hepatitis B (HBV) or hepatitis C (HCV) infection including hepatitis B surface antigen and hepatitis C antigen positive participants with or without abnormal liver enzymes (for SAD and MAD).
7. Evidence of any of the following (for SAD and MAD):

   1. creatinine ≥ 1.5 × ULN, or estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m^2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula at screening
   2. current hyper- or hypocalcemia, defined as albumin-adjusted serum calcium outside the normal range
   3. known intolerance to calcium supplements
   4. malignancy within the last 5 years, etc.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-01-13 (Actual); Study Completion 2024-01-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAE) in Part 1 (SAD). | Up to 85 days
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational product (IP), whether or not considered related to the IP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP.
Number of participants with clinically significant changes in total calcium (albumin-adjusted) in Part 1 (SAD). | Up to 85 days
  Serum calcium tested at Day 2, 4, 6, 15, 29, 85.
Number of participants with clinically significant changes in blood pressure in Part 1 (SAD). | Up to 85 days
  Systolic and diastolic blood pressure measured (mmHg) at all clinic visits (Day 1, 2, 3, 4, 5, 6, 8, 11, 15, 22, 29, 43, 57, 71, 85).
Number of participants with clinically significant changes in heart rate in Part 1 (SAD). | Up to 85 days
  Heart rate measured by electrocardiogram (ECG) on Day 1, 2, 4, 6, 15, 29, 85.
Number of participants with clinically significant changes in QTcF in Part 1 (SAD). | Up to 85 days
  QTcF (QT interval corrected for heart rate using Fridericia's formula) measured by electrocardiogram (ECG) on Day 1, 2, 4, 6, 15, 29, 43, 57, 71, 85.
Number of participants with treatment-emergent adverse events (TEAE) in Part 2 (MAD). | Up to 169 days
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational product (IP), whether or not considered related to the IP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP.
Number of participants with clinically significant changes in total calcium (albumin-adjusted) in Part 2 (MAD). | Up to 169 days
  Serum calcium tested at Day 2, 8, 15, 29, 36, 57, 64, 85, 169.
Number of participants with clinically significant changes in blood pressure in Part 2 (MAD). | Up to 169 days
  Systolic and diastolic blood pressure measured (mmHg) at all clinic visits (Day 1, 2, 4, 6, 8, 15, 22, 29, 36, 43, 57, 58, 60, 62, 64, 71, 78, 85, 99, 113, 127, 141, 155, 169).
Number of participants with clinically significant changes in heart rate in Part 2 (MAD). | Up to day 169
  Heart rate measured by electrocardiogram (ECG) on Day 1, 2, 4, 15, 29, 36, 57, 64, 85, 169.
Number of participants with clinically significant changes in QTcF in Part 2 (MAD). | Up to day 169
  QTcF (QT interval corrected for heart rate using Fridericia's formula) measured by electrocardiogram (ECG) on Day 1, 2, 4, 15, 29, 36, 57, 64, 85, 169.

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of AGA2118 | Part 1 (SAD): up to day 85; Part 2 (MAD) up to day 169
  Maximum concentration of AGA2118 after dosing.
Time to maximum concentration (Tmax) of AGA2118 | Part 1 (SAD): up to day 85; Part 2 (MAD) up to day 169
  Time to maximum concentration of AGA2118 after dosing.
Area under the concentration time curve (AUC) | Part 1 (SAD): up to day 85; Part 2 (MAD) up to day 169
  Definite integral of the curve describing the variation of AGA2118 in blood as a function of time.
Terminal elimination half-life (t1/2) | Part 1 (SAD): up to day 85; Part 2 (MAD) up to day 169
  Time it takes for maximum concentration to half of maximum concentration of AGA2118.

CONTACTS AND LOCATIONS:
Overall Officials: Angitia Medical Director, Study Director — Angitia Incorporated Limited
Locations (2):
- Australia (2):
  - Q-Pharm Pty Ltd, Brisbane, Queensland
  - Nucleus Network Pty Ltd., Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No